CLINICAL TRIAL: NCT02502435
Title: Exploratory Phase I Study to Define Plasma Fatty Acid Oscillations in Patients With Night Eating Syndrome Compared to Healthy Volunteers.
Brief Title: Human Plasma Fatty Acid Oscillations
Status: Suspended | Type: Observational
Why Stopped: COVID-19
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Carsten Skarke, MD, Research Assistant Professor, University of Pennsylvania
Other Study IDs: 819453
Record Dates: First submitted 2015-07-02; First posted 2015-07-20 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Nocturnal Eating-Drinking Syndrome; Healthy
MeSH Terms: conditions — Dyssomnias | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genetic analysis will be performed using High Throughput Sequencing (HTS) technology.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Night-Eating Syndrome: Individuals diagnosed with Night Eating Syndrome (NES); 18-65 years of age; eating 30% of their caloric intake after dinner with nocturnal awakenings to eat at a frequency of ≥ 5 times per week
  Interventions: Other: Observation
- Matched Healthy Controls: Healthy volunteers; 18-65 years of age; eating <25% of their caloric intake after dinner; no nocturnal ingestions
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observational study

SUMMARY:
This study wishes to look at the 24-hour rhythm of certain fats in the blood stream. Recent studies in animals and healthy participants suggest that unusual eating habits may be connected to a change in the 24-hour rhythm of the blood fats the investigators wish to measure. The investigators will ask persons suffering from night eating syndrome, a condition where people eat additional meals throughout the night, to participate in this study. Healthy volunteers who are of the same age and gender, and have a comparable body-mass-index, a number calculated from a person's weight and height, will also be asked to participate.

The aim is to learn how the 24-hour rhythm of the blood fats the investigators measure differs between the persons experiencing the night eating episodes and persons who do not.

DETAILED DESCRIPTION:
A disease mechanism driving the clinical symptomology of the Night Eating Syndrome (NES) may be a metabolome, polyunsaturated fatty acids in particular, disrupted in its oscillations throughout the course of day and night. Blood and stool samples will be repeatedly taken during a 3-night/2-day protocol from NES patients and healthy controls with lights dimmed to 20 lux and time cues removed. Body core temperature and physical activity during the study will be monitored continuously.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must be in good health as based on medical history, physical examination, vital signs, and laboratory tests as deemed by PI, BMI of 27-32;
* Volunteers are capable of giving informed consent;
* 18-65 years of age;
* Non-smoking; and
* Non-pregnant, female subjects must consent to a urine pregnancy test.
* Control subjects eat less than 25% of their caloric intake after dinner without nocturnal ingestions;
* NES patients have to meet both of the criteria for nocturnal ingestions and evening hyperphagia; eat 30% of their caloric intake after dinner with nocturnal wake ups to eat at a frequency of ≥ 5 times per week

Exclusion Criteria:

* Recent travel across time zones (within the past month);
* Planned travel across time zones during the planned study activities;
* Volunteers with irregular work hours, e.g. night shifts or swing shift schedule;
* Subjects, who have received an experimental drug, used an experimental medical device within 30 days prior to screening, or who gave a blood donation of ≥ one pint within 8 weeks prior to screening;
* Subjects with any abnormal laboratory value or physical finding that according to the investigator may interfere with interpretation of the study results, be indicative of an underlying disease state, or compromise the safety of a potential subject;
* Diagnosis of severe depression, lifetime diagnosis of bipolar disorder or any psychotic disorder;
* Prescription and non-prescription (OTC) medication; medication with psychotropics (including hypnotics);
* Actively participating in a weight loss diet or program;
* Diagnosed with a different eating disorder; and lack of awareness of the night eating episodes (to differentiate from nocturnal sleep-related eating disorder, in which nocturnal eating is accompanied by a lack of awareness at the time and amnesia for the behavior the following day.)

Exclusionary Medications and Substances

* Subjects who have taken medications including antibiotics 2 weeks prior to the start of the study and throughout the study deemed by the investigator to interfere with the measurement of the study. Birth control pills are acceptable and will not be excluded;
* Subjects who have taken aspirin or aspirin containing products for the 2 weeks prior to the start of the study and throughout the study;
* Subjects who have taken acetaminophen, NSAIDS, COX-2 inhibitors (OTC or prescription) for 1 week prior to the start of the study and throughout the study;
* Subjects who are currently consuming any type of tobacco product(s);
* Use of recreational drugs within the last 6 months;
* Subjects who consume high doses of antioxidant vitamins daily (vitamin C > 1000mg, Vitamin E > 400 IU, Beta Carotene > 1000IU, Vitamin A > 5000IU, Selenium > 200mcg, Folic Acid > 1mg) for the 2 weeks prior to the start of the study and throughout the study;
* Subjects who consume caffeine or high fat food 72 hours prior to the start of each study visit;
* Subjects need to abstain from alcohol consumption for 72 hours prior to the start of each study visit and throughout the active study.

Contraindications for the use of ingestible Temperature Sensors:

Screening for the contraindications listed below will occur during the physical and medical examination by a registered CTRC nurse or nurse practitioner:

* In any patient whose body weight is less than eighty (80) pounds.
* In the presence of any known or suspected obstructive disease of the gastrointestinal tract, including but not limited to diverticulitis and inflammatory bowel disease.
* In any patient exhibiting or having a history of disorders or impairment of the gag reflex.
* In any patient with previous gastrointestinal surgery.
* In any patient having fenilization of the esophagus.
* In any patient who might undergo Nuclear Magnetic Resonance (NMR) or MRI scanning during the period that the CorTemp® Disposable Temperature Sensor is within the body.
* In any patient with hypo motility disorders of the gastrointestinal tract including but not limited to Ileus.
* In any patient having a cardiac pacemaker or other implanted electro medical device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Night-Eating Syndrome: Participants have to meet both of the criteria for nocturnal ingestions and evening hyperphagia; eat 30% of their caloric intake after dinner with nocturnal wake ups to eat at a frequency of ≥ 5 times per week.
  Matching healthy participants: Participantswill be matched to a patient with Night-Eating Syndrome by gender, age and BMI.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Plasma fatty acids | 64 hours
  [% total fatty acid pool]

SECONDARY OUTCOMES:
Blood metabolite concentrations | 64 hours
  [uM]
Core body temperature | 64 hours
  [degrees C]
Bacterial taxa | 64 hours
  The proportions of the genus "Firmicutes Streptococcus" differences between mornings (0, 24, 48 hours) versus evenings (12, 36 hours) in microbiota collected by oral swabs from the left and right cheek.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Paschos, PhD, Principal Investigator — University of Pennsylvania; Kelly C Allison, PhD, Principal Investigator — University of Pennsylvania; Garret A FitzGerald, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Institute for Translational Medicine and Therapeutics (ITMAT), University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Center for Weight and Eating Disorders — http://www.med.upenn.edu/weight/allison.shtml
- See also: FitzGerald Lab — http://www.med.upenn.edu/fitzgeraldlab/